CLINICAL TRIAL: NCT06532721
Title: Child Development and Genetic Biomarkers(II): Gene Verification and Data Integration
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GENE-CGMH 2023 (DD)
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-05

CONDITIONS: Developmental Disabilities
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- developmental disabilities group: this group recruited children with developmental disabilities
- typical developmental group: This regoup recruited children with typical development

SUMMARY:
The aims of the study include (1) identifying genes associated with child development and developmental delay in Taiwan (2) comparing the differences and similarities between genetic biomarkers of development and developmental delay for children in Taiwan and children from other countries (3) employing precision medicine as the method for genetic screening or test and (4) tracking children's biological, psychological and social adjustment, especially for those who have early-onset developmental delay.

DETAILED DESCRIPTION:
The aims of the study include (1) identifying genes associated with child development and developmental delay in Taiwan (2) comparing the differences and similarities between genetic biomarkers of development and developmental delay for children in Taiwan and children from other countries (3) employing precision medicine as the method for genetic screening or test and (4) tracking children's biological, psychological and social adjustment, especially for those who have early-onset developmental delay.

The study will be completed in two phases over three years and will enroll a total of 475 0~40-year-old participants. In the first phase, we will recruit 380 participants. Including 50 participants with typical development, 300 participants with developmental delay and 30 parents to whom have children with severe DD. Then, their genetic data will be compared with genetic data of Chang Gung Hospital and the National Center for Genome Medicine, expect to preliminary find genes associated with child language development. At the same time, 20-30 children with severe developmental delay or have family history of developmental delay will be selected as a pilot study, using whole-exome sequencing (WES) to find other genes associated with development. If the gene deficiency was found in the children, we will invite his or her parents to do WES. In the second phase, we will establish a gene panel according to the genes identified in the previous stage and recruit 95 children with developmental delay to test the gene panel prospectively. The long-term goal of this study is to establish a pioneer study for children

ELIGIBILITY:
Inclusion Criteria:

* Consent signing
* 0-40 years old
* Typical development or developmental disabilities

Exclusion Criteria:

* Central Nervous disease
* Neuromuscular disease
* Congenital disease
* Sensory disorder such as blindness or hearing impairment

Max Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 475 participants with developmental disabilities and 50 healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 525 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Wechsler Preschool and Primary Scale of Intelligence | initial assessment
  Assess participant's intelligence.
  Verbal Comprehension Index:
  * Minimum Value :50
  * Maximum Value : 150
  * Interpretation : Higher score indicate better verbal reasoning, concept formation, and verbal comprehension abilities.
  Visual Spatial Index:
  * Minimum Value :50
  * Maximum Value : 150
  * Interpretation : Higher score indicate better visual-spatial reasoning and problem solving skills.
  Fluid Reasoning Index:
  * Minimum Value :50
  * Maximum Value : 150
  * Interpretation : Higher score indicate stronger abilities in abstract reasoning and problem solving skills.
  Working Memory Index:
  * Minimum Value :50
  * Maximum Value : 150
  * Interpretation : Higher score indicate better working memory, whic
Test of Nonverbal Intelligence-Fourth Edition | initial assessment
  assess participant's intelligence.
Cantab | initial assessment
  Assess participant's cognitive function
  Motor Screening Task:
  * Assess basic motor control and response to visual stimuli.
  * Measurement: Reaction time and movement time.
  * Faster response times indicate better motor function. Slower time suggest motor impairments or difficulties in visual processing.
  Paired Associates Learning:
  * Tests visual memory and new learning.
  * Measurement: Number of errors made during the task.
  * Higher error rated indicate poorer memory performance. Lower error rates suggest better visual memory and associative learning.
  Spatial Working Memory:
  * Assess the ability to retain and manipulate spatial information
  * Measurement: Number of errors and strategy scores.
  * Fewer errors and better strategy scores indicate better spatial working memory.
  Rapid Visual Information Processing:
  * Evaluates sustained attention and vigilance.
  * Measurements: Detection targets sequences within rapidly presented digits.
  * Higher hit rates and lower false
Peabody Picture Vocabulary Test-Revised | initial assessment
  Assess participant's language function.
Clancy Behavior Scale | initial assessment
  Help identifying autism symptoms.
  The scale covers multiple behavioral domains such as aggression, anxiety, social skills, attention and hyperactivity.
  The scale is administered as a questionnaire where parents, or caregivers rate the frequency and intensity of specific behaviors shown by the children. Responses are given on a Likert scale of 3.
  Minimum value: The scale's scoring system ranges from 0 (indicating no problematic behavior) to higher value of 2, depending on the number of items and the severity of the behavior assessed.
  Maximum value: The upper end of the scale is determined by the total number of items and the scoring format.
  Higher scores typically indicate more frequent or severe behavioral issues, while lower scores suggest fewer or less sever issues.
Swanson, Nolan, and Pelham, version IV | initial assessment
  screen ADHD symptoms.
The Berry-Buktenica Developmental Test of Visual-Motor Integration | initial assessment
  Assess participant's motor function.
Comprehensive Developmental Inventory for Infants and Toddlers | initial assessment
  Assess participant's general development.
Functional Independence Measure for Children | initial assessment
  Assess functional abilities of children and adolescents
  The WeeFIM includes three primary domains:
  * Self-care: Assesses the ability to perform basic self-care tasks independently.
  * Mobility: Measures the ability to move from one place to another and perform transfer.
  * Cognition: Evaluates cognitive abilities related to communication, social skills, and problem-solving.
  Rating scale: Each of the 18 items is rated on a 7-point scale based on the level of independence.
  Minimum Score: 18 (indicating complete dependence across all items) Maximum Score: 126 (indicating complete independence across all items)
  Higher score indicate greater functional independence, meaning the child requires less assistance to perform daily activities.
  Lower score indicate greater dependence, suggesting the child requires more assistance or is unable to perform certain tasks independently.
Assessment of Preschool Children's Participation | initial assessment
  Assess participant's participation in every day tasks.
Children Assessment of Participation and Enjoyment and Preferences for Activity of Children | initial assessment
  Assess participant's participation in every day tasks.
  The CAPE and PAC are designed for children and adolescents aged 6 to 21 years.
  Both tools are typically administered through structured questionnaires or interviews, either in paper form or electronically.
  CAPE: Helps identify areas where a child may be under-participating, guiding interventions to encourage greater engagement in a wider variety of activities.
  PAC: Provides insight into activities the child is interested in but may not currently participate in, helping to tailor activities to their preferences.
  Scoring:
  CAPE: Higher diversity and intensity scores indicate more varied and frequent participation. Higher enjoyment scores indicate greater pleasure derived from activities.
  PAC: Higher scores indicate a stronger preference for specific activities.
PedsQL TM | initial assessment
  Assess participant's quality of life.
  Core Scales:
  * Physical Functioning: Assesses difficulties with physical activities, such as walking, running, and participating in sports.
  * Emotional Functioning: Evaluates feelings of sadness, worry, and anger, as well as overall emotional well-being.
  * Social Functioning: Measures interactions with peers, the ability to make friends, and feelings or being excluded or bullied.
  * School Functioning: Assesses difficulties in paying attention in class, missing school due to illness, and keeping up with schoolwork.
  The PedsQl uses a 5-point likert scale for responses.
  Higher score indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: ChiaLing Chen, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No